CLINICAL TRIAL: NCT03822728
Title: Postoperative Facial Weakness in Parotidectomy for Deep Seated Parotid Tumor With or Without Intra-parotid Facial Nerve Imaging (3D Double-Echo Steady-State With Water Excitation MRI Imaging)
Brief Title: Intra-parotid Facial Nerve Imaging in Parotidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Han-Sin Jeong, Professor, Samsung Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-07-084
Record Dates: First submitted 2019-01-29; First posted 2019-01-30 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Parotid Tumors; Facial Nerve Paresis
MeSH Terms: conditions — Parotid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Without 3D-DESS MRI (No Intervention): As for deep seated tumors in preoperative CT or US (or tumors in both superficial and deep parotid glands), the patients will undergo surgery without 3D-DESS MRI (currently routine practice).
- With 3D-DESS MRI (Experimental): As for deep seated tumors in preoperative CT or US (or tumors in both superficial and deep parotid glands), preoperative 3D-DESS MRI will be additionally performed to delineate the intra-parotid facial nerve.
  Interventions: Diagnostic Test: 3D-DESS MRI (3 dimensional double echo steady state MRI)

INTERVENTIONS:
Diagnostic Test: 3D-DESS MRI (3 dimensional double echo steady state MRI) — 3D-DESS MRI has been reported useful for the intra-parotid facial nerve imaging. It can provide information about the anatomical relationship between the tumor and the facial nerve in the parotid gland.
  Arms: With 3D-DESS MRI

SUMMARY:
In this study, the investigators will evaluate the clinical usefulness of 3 dimensional double echo steady state MRI (3D-DESS MRI) for functional preservation of the facial nerve during parotidectomy. Preoperative 3D-DESS MRI imaging can provide information about the anatomical relationship between the tumor and the facial nerve in the parotid gland.

Because the risk of postoperative facial weakness is relatively high in the deep-seated parotid tumors, the investigators will exclude the patients with the superficial parotid tumors (determined by preoperative CT or US) and only include the patients with deep seated parotid tumors in this trial.

The main outcome of our study is the incidence of immediate postoperative facial weakness, and the secondary outcome is the incidence of facial weakness at postoperative 6 months.

DETAILED DESCRIPTION:
Surgical removal of tumors arising from the parotid gland (benign or malignant) is treatment of choice. However, the most detrimental complication of parotidectomy is facial weakness or facial nerve palsy, because the facial nerve crosses in the mid-portion of the parotid gland.

Numerous studies indicated the incidence of temporary facial weakness as 5-45% and permanent facial palsy as 0-15% after parotidectomy. To reduce this complication, the investigators will apply the modern technique of MRI imaging to inform the anatomical relationship between the tumor and the facial nerve within the parotid gland preoperatively. Three dimensional double echo steady state MRI imaging (3D-DESS MRI) has been reported useful for the intra-parotid facial nerve imaging.

Thus, the investigators will evaluate the clinical usefulness of 3D-DESS MRI for functional preservation of the facial nerve during parotidectomy. Preoperative 3D-DESS MRI imaging can provide information about the anatomical relationship between the tumor and the facial nerve in the parotid gland.

In the retrospective series, the investigators found that there were 25.6% temporary facial weakness and 10.3% permanent (> 6 months) facial weakness after parotidectomy for deep-seated parotid tumors (plus tumors located in both deep and superficial parotid gland); whereas 6.7% and 3.6% facial weakness respectively for superficially located parotid tumors. Because the risk of postoperative facial weakness is relatively high in the deep-seated parotid tumors, the investigators will exclude the patients with the superficial parotid tumors (determined by preoperative CT or US) and only include the patients with deep seated parotid tumors in this trial.

The main outcome of our study is the incidence of immediate postoperative facial weakness, and the secondary outcome is the incidence of facial weakness at postoperative 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Parotid tumors subject to the surgery (parotidectomy)
* Parotid deep lobe tumors or tumor located in both superficial and deep parotid glands (Tumor medial to the facial nerve line, a line connecting the lateral border of mandible and the posterior belly of digastric muscle on CT scans or tumors crossing the facial nerve line on CT scans)
* Benign or malignant tumors
* Any size of parotid tumors

Exclusion Criteria:

* Superficially located parotid tumor on CT or US (Tumor lateral to the facial nerve line, a line connecting the lateral border of mandible and the posterior belly of digastric muscle on CT scans)
* Previous parotid surgery in the affected parotid gland (Revision parotid surgery)
* Preoperative facial nerve palsy
* Cases with the facial nerve sacrifice during surgery for oncological purpose (malignancy)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Immediate postoperative facial weakness | Postoperative day 1
  Evaluation of facial function using Facial palsy grading system, immediately after parotidectomy.
  Measures: House-Brackmann Facial Nerve Grading System (1: Normal, 2: Mild dysfunction, 3: Moderately dysfunction, 4: Moderately severe dysfunction, 5: Severe dysfunction, 6: Total paralysis)

SECONDARY OUTCOMES:
Permanent postoperative facial weakness | Postoperative 6 months
  Evaluation of facial function using Facial palsy grading system, at 6 months after parotidectomy.
  Measures: House-Brackmann Facial Nerve Grading System (1: Normal, 2: Mild dysfunction, 3: Moderately dysfunction, 4: Moderately severe dysfunction, 5: Severe dysfunction, 6: Total paralysis)

CONTACTS AND LOCATIONS:
Overall Officials: Han-Sin Jeong, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
The investigators will make our participant data available to other researchers after completion of this study.

REFERENCES:
- [Background] Qin Y, Zhang J, Li P, Wang Y. 3D double-echo steady-state with water excitation MR imaging of the intraparotid facial nerve at 1.5T: a pilot study. AJNR Am J Neuroradiol. 2011 Aug;32(7):1167-72. doi: 10.3174/ajnr.A2480. Epub 2011 May 12. PMID 21566007